CLINICAL TRIAL: NCT00245661
Title: Effects of Temazepam on Dyspnea, Gas Exchange and Sleep Quality in Chronic Obstructive Pulmonary Disease.
Brief Title: Effects of Temazepam in Patients With Chronic Pulmonary Obstructive Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LTC-346/050905/Stege
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; respiratory; sleep quality; temazepam; dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders; Dyspnea | interventions — Temazepam

INTERVENTIONS:
Drug: Temazepam

SUMMARY:
The purpose of this study is to evaluate the effects of temazepam during sleep and in daytime on dyspnea, gas exchange and sleep quality in patients with chronic obstructive pulmonary disease.

The study hypothesis is that temazepam does not produce any adverse respiratory effects during sleep in patients with COPD. In contrast, it may result in an beneficiary effect because it positively affects the sleep quality and sleep structure which may result in more alertness and less daytime sleepiness and less dyspnea during the day.

DETAILED DESCRIPTION:
Rationale: More than 50% of patients with chronic obstructive pulmonary disease (COPD) have sleep complaints characterised by longer latency to falling asleep, more frequent arousals and awakenings, generalised insomnia and/or excessive daytime sleepiness. Sleep disturbance seems to be more severe with advancing disease and substantially reduces patients' quality of life. The sleep complaints are due to dyspnea, chronic cough, sputum production, hypoxaemia and hypercapnia during the night. One of the available therapies for these patients is the prescription of hypnotics (like benzodiazepines). However, it is thought that in patients with COPD sleep medication may produce adverse respiratory effects due to suppression of the cerebral respiratory drive. In our practice, we never encounter any adverse respiratory effect of an hypnotic in patients with COPD. There have been several trials in COPD patients studying these potentially adverse effects. The results of these studies are inconsistent, relative older hypnotics are used and there are several methodological limitations. Furthermore, in none of these studies transcutaneous PCO2 or PO2 was monitored. Temazepam is nowadays the sedative of first choice in the medical treatment of sleep complaints.

Aim: primary: studying the effects of temazepam on the respiratory function during daytime and at night in patients with severe COPD. Secondary: studying the effects of temazepam on the sleep quality and sleep structure and on the objective and subjective sleepiness during daytime and at night in patients with COPD.

Study design: double blind, placebo-controlled, cross-over randomised clinical trial.

Treatment: 10 mg temazepam or placebo during seven consecutive nights.

Endpoints: Primary: difference in PtcCO2, PtcO2 and oxygen saturation during sleep after 1 week temazepam compared to placebo. Secondary: Respiratory Disturbance Index, Desaturation Index and Hypercapnic Ventilatory Response, percentage REM/nREM-sleep and total effective sleep time, Multiple Sleep Latency Test and the Epworth Sleeping Score.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD, GOLD 3 or 4
* having subjective sleeping problems

  * longer latency to falling asleep
  * frequent arousals
  * excessive daytime sleepiness
* clinical stable health for minimally 6 weeks

Exclusion Criteria:

* usage of some sort of medication that influences sleep in any kind of way (like benzodiazepines, barbiturates, opiates, amfetamines) which can not be discontinued during the study period
* alcohol abuse
* hospitalisation 6 weeks or shorter before enrollment in the study
* hyperreactivity / allergy to benzodiazepines
* history of benzodiazepine-dependence
* myasthenia gravis
* obstructive sleep apnea syndrome (OSAS)
* severe liver failure
* age under 18 years
* participation in another study less than 6 weeks before enrollment
* COPD exacerbation less than 6 weeks before enrollment
* usage of oxygen supplementation at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2005-10; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
transcutaneous PCO2
transcutaneous PO2
Oxygen saturation

SECONDARY OUTCOMES:
Respiratory Disturbance Index
Desaturation Index
MSLT
arterial PO2
arterial PCO2
Hypercapnic Ventilatory Response
total sleeping time
sleep latency
percentage REM- and nREM-sleep of total sleep time
number of arousals
number of apneas during sleep
number of hypopneas during sleep
Epworth Sleeping Score
Dyspnea Visual Analog Score

CONTACTS AND LOCATIONS:
Overall Officials: Gerben Stege, MD, Principal Investigator — Rijnstate Hospital; Peter J de Bruijn, MD, Study Director — Rijnstate Hospital; Richard PN Dekhuijzen, Prof. PhD MD, Study Director — UMC St. Radboud; Frank JJ van den Elshout, PhD MD, Study Director — Rijnstate Hospital; Yvonne F Heijdra, PhD MD, Study Director — UMC St. Radboud; Marjo JT van de Ven, PhD MD, Study Director — Rijnstate Hospital; Petra JE Vos, PhD MD, Study Chair — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Derived] Stege G, Heijdra YF, van den Elshout FJ, van de Ven MJ, de Bruijn PJ, van Sorge AA, Dekhuijzen PN, Vos PJ. Temazepam 10mg does not affect breathing and gas exchange in patients with severe normocapnic COPD. Respir Med. 2010 Apr;104(4):518-24. doi: 10.1016/j.rmed.2009.10.022. Epub 2009 Nov 12. PMID 19910177
- See also: sponsor's web site — http://www.alysis.nl/site/index_html